CLINICAL TRIAL: NCT00690547
Title: Force Enhancement of m. Quadriceps Femoris During and After Excentric Muscle Activity in Vivo by Maximal and Sub-maximal Deliberately Activation.
Brief Title: Force Enhancement of Musculus Quadriceps Femoris During and After Excentric Muscle Activity in Vivo
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: German Research Foundation (Other)
Responsible Party: Prof. Dr. Ansgar Schwirtz, Technical University of Munich, Department of Biomechanics in Sports
Other Study IDs: DFG27112007
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: Muscle Quadriceps Femoris; Healthy
Keywords: Functionality; Deliberately; Activated; Quadriceps; Femoris; During; After; Active; Extension
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Test Group
  Interventions: Other: muscle activation

INTERVENTIONS:
Other: muscle activation — activation of the muscle quadriceps femoris

SUMMARY:
Force enhancement (FE) describes the phenomenon of strength potentialization of a muscle cell or the complete muscle during and after active extension compared to the strength of an isometric contraction with same muscle length. The underlying physiological mechanism of this phenomenon is not completely known today. In vitro trials indicate that the interaction of an active and a passive component on the cellular level are responsible for the higher strength measurements. So far FE could be shown in vitro and in vivo on muscle fibers and small human muscles. Further research is needed for verification of the existence of FE in voluntary motor activity in everyday life. In order to approach this objective the investigators will scrutinize the functionality of the deliberately activated musculus (m) quadriceps femoris during and after active extension on the basis of in vivo studies.

DETAILED DESCRIPTION:
The research proposal is resubmitted with no amendments made regarding content.

ELIGIBILITY:
Inclusion Criteria:

* Males without previous muscular or neurophysiological diseases
* Age between 20 and 40 years

Exclusion Criteria:

* Previous muscular or neurophysiological diseases

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: males without previous muscular or neurophysiological diseases at an age between 20 and 40 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Identification of a potential Force enhancement by complex muscle activity with a high relevance for everyday life, for example more agile leg stretching (knee bend). | 12 months

SECONDARY OUTCOMES:
Evidence of existence of the force enhancement by deliberately activated, great human muscle by sub-maximal activation | 12 months
Correlation between typ of muscle fiber and force enhancement in vivo | 12 months
Analysis of the alternation of length of the muscle fiber during and after excentric extension for the differentiated explanation of in vivo mechanism excentric and post-excentric strength | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ansgar Schmirtz, Prof. Dr., Principal Investigator — Technical University of Munich, Department of Biomechanics in Sports
Locations (1):
- Technical University of Munich, Department of Biomechanics in Sports, Munich, Germany